CLINICAL TRIAL: NCT04427085
Title: Optic Nerve Sheath Diameter Between Obese and Non-obese Patients Undergoing Laparoscopic Gynecological Surgery
Brief Title: Changes of Optic Nerve Sheath Diameter Between Obese and Non-obese Patients Undergoing Laparoscopic Gynecological Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Associate professor, SMG-SNU Boramae Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 20421
Record Dates: First submitted 2020-04-22; First posted 2020-06-11 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Optic Nerve Sheath Diameter

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obese group (Experimental): body mass index≥ 30 kg/m2
  Interventions: Other: Ultrasound assessment of optic nerve sheath diameter
- Non-obese group (Active Comparator): BMI < 30 kg/m2
  Interventions: Other: Ultrasound assessment of optic nerve sheath diameter

INTERVENTIONS:
Other: Ultrasound assessment of optic nerve sheath diameter — Using ultrasonography, optic nerve sheath diameter is measured during perioperative period.

SUMMARY:
This study aims to compare the change of optic nerve sheath diameter in obese and non-obese patients undergoing laparoscopic gynecological surgery in a steep Trendelenburg position.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic gynecological surgery

Exclusion Criteria:

* Ophthalmic diseases
* Previous history of ophthalmic surgery.
* Neurological disorders
* History of head surgery.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
Optic nerve sheath diameter | 30 minutes after pneuroperitoneum in the Trendelenburg position
  Using ultrasonography, optic nerve sheath diameter is measured.

SECONDARY OUTCOMES:
Optic nerve sheath diameter | 15 minutes after pneuroperitoneum in the Trendelenburg position
  Using ultrasonography, optic nerve sheath diameter is measured.
Optic nerve sheath diameter | 60 minutes after pneuroperitoneum in the Trendelenburg position
  Using ultrasonography, optic nerve sheath diameter is measured.
Optic nerve sheath diameter | 10 minutes after release of pneumoperitoneum and return to the supine position
  Using ultrasonography, optic nerve sheath diameter is measured.
Optic nerve sheath diameter | At 1 hour after completion of surgery
  Using ultrasonography, optic nerve sheath diameter is measured.
Optic nerve sheath diameter | At 24 hours after completion of surgery
  Using ultrasonography, optic nerve sheath diameter is measured.
Nausea and vomiting | At 1 hour after completion of surgery
  The presence and severity of nausea and vomiting is evaluated.
Headache | At 1 hour after completion of surgery
  The presence and severity of headache is evaluated.
Nausea and vomiting | At 24 hours after completion of surgery
  The presence and severity of nausea and vomiting is evaluated.
Headache | At 24 hours after completion of surgery
  The presence and severity of headache is evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, South Korea